CLINICAL TRIAL: NCT01013207
Title: Assessment of the Compliance and Usability of the Nexus (S9) CPAP System in Sleep Disordered Breathing
Brief Title: Nexus Compliance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Klaus Schindhelm: Professor, Graduate School of Biomedical Engineering, UNSW, ResMed
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MA051109
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Results first posted 2010-09-01 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: CPAP compliance
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nexus (S9) CPAP device (Experimental): Fifty subjects with obstructive sleep apnea (OSA), established on CPAP therapy (≥ 6 months) were recruited into this study. These patients use their CPAP device every night while sleeping to treat their OSA.
  Nexus (S9) is a new CPAP device with improved humidification system (heated tube and climate control), reduced noise, improved comfort of breathing and new user interface. During the study, patients will use this CPAP every night in place of their own CPAP for a period of 4 weeks. Compliance data from the Nexus will then be compared to the patient's usual CPAP pre trialling Nexus and post trialling Nexus.
  Interventions: Device: CPAP Pre Nexus (S9); Device: Nexus (S9); Device: CPAP Post Nexus (S9)

INTERVENTIONS:
Device: CPAP Pre Nexus (S9) — This is the patient's own CPAP prior to trialling the Nexus (S9). 4 weeks of data will be downloaded from this device and compared to 4 weeks using Nexus (S9), and 4 weeks usage post trialling Nexus (S9)
  Other Names: Patient's own CPAP
Device: Nexus (S9) — The patient will use the new Nexus (S9) CPAP for four weeks in place of their usual CPAP every night when they sleep to treat their OSA. Compliance data will be compared between four weeks on this device to the last four weeks on their current device (CPAP Pre S9). After using the Nexus (S9) CPAP for four weeks, participants will return to their current device for four weeks. Data from this post-trial period will be compared with both the Nexus (S9) four weeks, and the four weeks pre Nexus (S9) usage.
  Other Names: S9 AutoSet
Device: CPAP Post Nexus (S9) — After trialling the Nexus (S9) for four weeks, patients will return to their usual CPAP. Data from the patient's usual CPAP for four weeks will be compared to data while using the Nexus (S9), and data from the patient's usual device pre trialling S9 (CPAP Pre Nexus)
  Other Names: Patient's own CPAP

SUMMARY:
Obstructive sleep apnoea (OSA) is characterised by a partial or complete collapse of the upper airway during sleep. The treatment of choice for OSA is Continuous Positive Airway Pressure (CPAP). CPAP acts as a positive airway splint, delivering a fixed positive airway pressure to the upper airway via a tube and mask. Humidification is used during CPAP therapy to improve the comfort of the delivered air and to alleviate nasal dryness/congestion.

The latest design of a CPAP device, known as Nexus (S9), encompasses new features including an improved humidification system (heated tube and climate control), reduced noise, improved comfort of breathing, and a new user interface.

This study will assess whether compliance on CPAP therapy is improved on the Nexus (S9) CPAP, and will assess the usability of the Nexus (S9) CPAP

DETAILED DESCRIPTION:
Obstructive Sleep Apnoea (OSA) is a condition characterised by the partial or complete collapse of the upper airway during sleep. OSA comprises a continuous spectrum of severity ranging from simple snoring and upper airway resistance through mild to severe symptomatic obstructive hypopnoea and apnoea. The prevalence of sleep disordered breathing in the adult population is 24% males and 9% for females. The prevalence of symptomatic OSA in the adult population has been estimated to be 4% in males and 2% in females. These patients demonstrate behavioural and neuropsychological consequences to varying degrees, including excessive daytime sleepiness, intellectual deterioration and depression. More serious consequences include arterial systemic hypertension, arterial pulmonary hypertension and heart disease.

The treatment of choice for OSA is Continuous Positive Airway Pressure (CPAP). CPAP acts as a positive airway splint, delivering a fixed positive airway pressure to the upper airway via a tube and mask. Humidification is used during CPAP therapy to improve comfort of the delivered air and alleviate nasal dryness/congestion.

Compliance with CPAP is a known issue which is affected by many things, including negative side effects and issues with the equipment. The most common complaints involve nasal dryness/congestion and noise from the machine.

The purpose of this study is to assess whether the improved humidification system, reduced noise, improved comfort of breathing and new user interface on the Nexus (S9) CPAP will improve compliance.

Aims:

1. To determine if compliance on the new Nexus (S9) CPAP is improved over the patient's usual CPAP
2. To assess the usability of the Nexus (S9) CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide written informed consent
* Patients who are using a ResMed mask system
* Patients who are at least 18 years of age
* Patients who use a ResMed CPAP device

Exclusion Criteria:

* Patients currently using Bilevel PAP
* Patients who are pregnant
* Patients who the researcher believes are unsuitable for inclusion because either:

  * they do not comprehend English
  * they are unable to provide written informed consent
  * they are physically unable to comply with the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schindhelm, PhD, Principal Investigator — ResMed
Locations (1):
- ResMed Sleep Reseach Centre, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Wimms AJ, Richards GN, Benjafield AV. Assessment of the impact on compliance of a new CPAP system in obstructive sleep apnea. Sleep Breath. 2013 Mar;17(1):69-76. doi: 10.1007/s11325-012-0651-0. PMID 22286779

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from ResMed Science Centre, Sydney, between November 2009 and March 2010
Period: CPAP Pre Nexus (S9)
Arm/Group | All Participants
Started | 50
Completed | 50
Not Completed | 0
Period: Nexus (S9)
Arm/Group | All Participants
Started | 50
Completed | 50
Not Completed | 0
Period: CPAP Post Nexus (S9)
Arm/Group | All Participants
Started | 50
Completed | 44
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 32
Region of Enrollment [Number; unit: participants]
  Australia | 50

OUTCOME MEASURES:

1. Primary Outcome: Compliance on CPAP
Description: Compliance on CPAP was measured as average daily usage
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | All Participants
Number analyzed (Participants) | 50
Hours
  CPAP Pre Nexus (S9) | 6.58 (1.95)
  Nexus (S9) | 7.07 (1.2)
  CPAP Post Nexus (S9) | 6.72 (1.2)

2. Secondary Outcome: Usability of the Nexus (S9) CPAP.
Description: The usability quesitonnaire was administered at the end of the 4 week trial of Nexus (S9). Usability was defined as ease of using the Nexus (S9) and overall satisfaction with the Nexus (S9) CPAP. The outcome measure was collected through 11 point Likert questionnaires, where 0 = very poor usability and 10 = excellent usability.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 50
Units on a scale | 9.48 (1.03)

ADVERSE EVENTS:
Time Frame: 2 months
Description: Adverse events were collected after 1 week, 1 month and 2 months from the beginning of the study. Adverse events were collected/ assessed through clinical interview. No adverse events were reported or observed during the study.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes